CLINICAL TRIAL: NCT04532294
Title: A First-in-Human, Randomized, Double-Blind, Placebo Controlled, Single Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of SARS-CoV-2 Neutralizing Antibody BGB-DXP593 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2/COVID-19) Neutralizing Antibody in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BGB-DXP593-101
Record Dates: First submitted 2020-08-27; First posted 2020-08-31 (Actual); Results first posted 2022-01-27 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BGB-DXP593: Dose Level A (Experimental): Participants will receive BGB-DXP593 10 mg/kg on Day 1
  Interventions: Drug: BGB DXP593
- BGB-DXP593: Dose Level B (Experimental): Participants will receive BGB-DXP593 30 mg/kg on Day 1
  Interventions: Drug: BGB DXP593
- Placebo (Experimental): Placebo to match (PTM) BGB-DXP593 on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGB DXP593 — Administered intravenously (IV) as specified in the treatment arm
  Arms: BGB-DXP593: Dose Level A; BGB-DXP593: Dose Level B
Drug: Placebo — Placebo to match BGB-DXP593
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to investigate the safety and tolerability of BGB-DXP593 administered intravenously as a single dose in healthy participants

ELIGIBILITY:
Key Inclusion Criteria :

1. Participants are in good general health as determined by the investigator or medically qualified designee, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring
2. Body weight ≥ 50 kg and body mass index (BMI) within the range 18 to 32 kg/m2 (inclusive) Note: BMI = weight [kg] / (height [m])
3. Negative serum IgG to the SARS-CoV-2
4. Negative for COVID-19 based on the nasopharyngeal or oropharyngeal swab with the method of real-time reverse transcription-polymerase chain reaction (rRT-PCR)

Key Exclusion Criteria:

1. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs, constituting a risk to the participant when taking the study drug; or interfering with the interpretation of data
2. Any history of a severe allergic reaction prior to enrollment that has a reasonable risk of recurrence during the study
3. Have a medical history of SARS infection
4. Any acute fever disease or infections
5. Any chronic or clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety or rights of the participant, including but not limited to: diabetes mellitus type I, chronic hepatitis; or clinically significant forms of: drug or alcohol abuse, asthma (except for childhood asthma), autoimmune disease, psychiatric disorders, or heart disease

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2021-02-13 (Actual); Study Completion 2021-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Principal Investigator — BeiGene
Locations (1):
- Q PHARM, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received a single intravenous dose of matching placebo
- BGB-DXP593 10 mg/kg: Participants received a single 10 milligrams/kilogram (mg/kg) intravenous dose of BGB-DXP593
- BGB-DXP593 30 mg/kg: Participants received a single 30 milligrams/kilogram (mg/kg) intravenous dose of BGB-DXP593
Period: Overall Study
Arm/Group | Placebo | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Started | 4 | 6 | 8
Completed | 4 | 6 | 5
Not Completed | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Participants Not Dosed | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS) : Includes all participants who received the study drug or placebo
Groups:
- BGB-DXP593 10 mg/kg: Participants received a single 10 mg/kg intravenous dose of BGB-DXP593
- BGB-DXP593 30 mg/kg: Participants received a single 30 mg/kg intravenous dose of BGB-DXP593
- Total: Total of all reporting groups
Arm/Group | Placebo | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg | Total
Number analyzed (Participants) | 4 | 6 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.0 (13.64) | 34.2 (16.46) | 39.7 (14.81) | 35.4 (14.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 2 | 5
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 4 | 6 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 1 | 0 | 1
  White | 4 | 5 | 5 | 14
  Other | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE is defined as an adverse event (AE) that had an onset date or a worsening in severity from baseline on or after the administration of study drug and up to 30 days after the dose of study drug
Time Frame: From the day of study drug administration until 30 days after dose (up to approximately 160 days)
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 4 | 6 | 6
Participants
  Participants with at least 1 TEAE | 4 | 4 | 4
  Participants with SAEs | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Vital Signs and Electrocardiograms
Description: Systolic and diastolic blood pressure, pulse rate, body temperature, and respiratory rate were measured. Descriptive statistics for ECG parameters (heart rate and QTcF interval) and changes from baseline were summarized
Time Frame: Up to approximately 160 days
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 4 | 6 | 6
Participants
  Participants with changes in vital signs | 0 | 0 | 0
  Participants with changes in ECG | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Clinically Relevant Changes in Laboratory Parameters
Description: Clinical laboratory values were evaluated for each laboratory parameter as applicable including hematology, serum chemistry and urinalysis.
Time Frame: Up to approximately 160 days
Population: Safety analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 4 | 6 | 6
Participants | 0 | 0 | 0

4. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion, 6 hrs. post-dose), Days 2, 3, 4, 5, 8, 15, 22, 29, 43, 57, 71, 85 and End of study visit (Up to approximately160 days)
Population: Pharmacokinetic (PK) Analysis Set includes all the participants who received the study drug and had any measurable concentration of study drug.
Measure: Median (Full Range); unit: μg/mL
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
μg/mL | 255.3 [213 to 328] | 667.0 [511 to 787]

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Infinity (AUCinf) of BGB-DXP593
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
day*μg/mL | 4168.8 [3565 to 6188] | 12422.6 [9095 to 15810]

6. Secondary Outcome: AUC From Time Zero to Time of Last Quantifiable Concentration (AUClast) of BGB-DXP593
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
day*μg/mL | 3964.6 [3388 to 5887] | 11434.2 [8912 to 15334]

7. Secondary Outcome: AUC From Time Zero to Day 29 (AUC0-29) of BGB-DXP593
Time Frame: Day 1 (pre-dose, End of Infusion, 6 hrs. post-dose), Days 2, 3, 4, 5, 8, 15, 22, and 29
Population: PK Analysis Set
Measure: Median (Full Range); unit: day*μg/mL
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
day*μg/mL | 2368.4 [2052 to 3489] | 6683.9 [5919 to 9022]

8. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of BGB-DXP593
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Median (Full Range); unit: hours
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
hours | 1.47 [1.3 to 7.0] | 3.67 [1.2 to 24.0]

9. Secondary Outcome: Terminal Half Life (t1/2) of BGB-DXP593
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Median (Full Range); unit: Day
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
Day | 26.60 [20.4 to 32.1] | 25.77 [20.7 to 29.1]

10. Secondary Outcome: Clearance (CL) of BGB-DXP593
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Median (Full Range); unit: Liters/Day
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
Liters/Day | 0.18 [0.1 to 0.2] | 0.19 [0.1 to 0.2]

11. Secondary Outcome: Volume of Distribution (Vz) of BGB-DXP593
Time Frame: as for outcome 4
Population: PK Analysis Set
Measure: Median (Full Range); unit: Liters
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
Liters | 6.54 [3.1 to 8.1] | 6.30 [5.7 to 9.4]

12. Secondary Outcome: Immunogenic Response to BGB-DXP593 as Assessed by the Detection of Antidrug Antibodies (ADA)
Time Frame: Up to approximately160 days
Population: The ADA Analysis Set includes all the participants who received the study drug and in whom both baseline ADA and at least 1 postbaseline ADA results are available
Measure: Count of Participants; unit: Participants
Arm/Group | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
Number analyzed (Participants) | 6 | 6
Participants
  Treatment Induced ADA | 1 | 0
  Neutralizing antibody (NAb) Positive | 0 | 0

ADVERSE EVENTS:
Time Frame: From the day of study drug administration until 30 days after dose (Up to approximately160 days)
Arm/Group | Placebo | BGB-DXP593 10 mg/kg | BGB-DXP593 30 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/6 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=4) | BGB-DXP593 10 mg/kg (N=6) | BGB-DXP593 30 mg/kg (N=6)
Headache (Nervous system disorders) | 2 | 2 | 2
Presyncope (Nervous system disorders) | 1 | 0 | 0
Catheter site pain (General disorders) | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Catheter site swelling (General disorders) | 0 | 1 | 0
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Catheter site bruise (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT04532294/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04532294/SAP_001.pdf